| | Clinical Investigational Plan Synopsis Study Name: Substrate-targeted Catheter Ablation to |
|---|---|
| | Treat Atrial Fibrillation Ver. 1.0 11MAR2015 |
| Clinical Investigational Plan Synopsis | |

| Title: | Substrate-Targeted Catheter Ablation to Treat Persistent Atrial Fibrillation |
|---|---|
| Acronym: | AF Substrate Mapping and Guided Ablation |
| Purpose: | Evaluate the feasibility of substrate-targeted catheter ablation to treat Persistent AF |
| Objectives: | Primary Objective |
| | • Assess acute and long-term outcome of patient-tailored substrate-targeted ablation (Substrate) plus modified circumferential pulmonary vein ablation (Substrate+mCPVA) versus modified circumferential pulmonary vein ablation alone (mCPVA) |
| | Secondary Objective |
| | <ul> <li>Map and characterize electrophysiological substrates during AF,<br/>including regular and fast activities, complex fractionated<br/>electrograms, wave front propagation directions, and fibrosis</li> </ul> |
| Endpoints: | Primary Endpoint |
| | Twelve-month clinical success rate defined as |
| | <ul> <li>Freedom from symptomatic AF off antiarrhythmic drug therapy<br/>assessed from the end of the 3 months blanking period to 12<br/>months following the ablation procedure, documented by<br/>implantable loop recorder (ILR) monitoring or trans-telephonic</li> </ul> |
| | (TT) ECG monitoring. |
| | Secondary Endpoint |
| | <ul> <li>Collect maps that identify substrates that could serve as mechanisms of AF maintenance, such as: <ul> <li>Areas with fast but regular activities</li> <li>Areas with consistent wave front propagation pattern</li> <li>Areas with low P-P voltage</li> <li>Areas with complex fractionated electrograms</li> </ul> </li> <li>Acute AF termination or significant AF cycle length slowing during RF application in ablation procedure</li> <li>Inducibility of AF by programmed stimuli at the end of the ablation procedure before and after administration of Isoproterenol</li> <li>Freedom from symptomatic atrial tachycardia and atrial flutter off antiarrhythmic drug therapy assessed from the end of the 3 months blanking period to 12 months following the ablation procedure, documented by ILR monitoring or TT ECG monitoring</li> <li>Freedom from asymptomatic AF, atrial tachycardia, and atrial flutter off antiarrhythmic drug therapy assessed from the end of the 3 months blanking period to 12 months following the ablation procedure, documented by ILR monitoring or TT ECG monitoring</li> </ul> |
| | <ul> <li>Need for a new ablation procedure</li> <li>Need to prescribe antiarrhythmic drugs after the blanking period</li> <li>AF burden measured by ILR at follow-up visits</li> </ul> |

| Treat Atrial Fibrillation Ver. 1.0 11MAR2015 Clinical Investigational Plan Synopsis | |
|---|---|
| | Study Name: Substrate-targeted Catheter Ablation to |
| | Clinical Investigational Plan Synopsis |

| Design: | Prospective, single center, randomized, single-blind, controlled, 2-arm parallel group trial in Milan, Italy (Pr. Pappone, Targeted Research Center) |
|---|---|
| | The total duration of the study is expected to be 24 months with ~12 months of enrollment. |
| | <ul> <li>Approximately 80 subjects suffering from persistent AF will be randomized in a 1:1 fashion to the following investigation arms: <ul> <li>Modified circumferential pulmonary vein ablation alone (mCPVA);</li> <li>Substrate-targeted ablation guided by AF substrate mapping, followed by completion of modified circumferential pulmonary vein ablation (Substrate+ mCPVA)</li> </ul> </li> </ul> |
| | <ul> <li>Ablate the areas that have fast and regular electrical<br/>activities, starting from the fastest cycle length (defined by<br/>Mean CL in the range of 120-250 milliseconds, and SD CL<br/>in the range of 1-30 milliseconds</li> </ul> |
| | Ablate the areas that have consistent rotational or focal propagation pattern (defined by conduction velocity vectors) |
| | <ul> <li>Ablate the areas that comprises the slow conduction zone<br/>of possible arrhythmia circuits</li> </ul> |
| | <ul> <li>If AF terminates during RF ablation, stimulation protocol will be used to examine if AF is re-inducible. If AF is re- inducible and physician decides to remap, mapping will be performed again for substrate-targeted ablation. If AF is not re-inducible, mCPVA will be completed</li> </ul> |
| | Subjects will be followed up at 3, 6, 12 months |
| Devices used: | Subjects will be followed up at 3, 6, 12 months. - EnSite <sup>TM</sup> Velocity <sup>TM</sup> mapping system (CE marked) TM A F H <sup>TM</sup> 1: (CF 1 1) |
| | <ul> <li>Inquiry<sup>TM</sup> AFocusII<sup>TM</sup> diagnostic catheter (CE marked)</li> <li>EnSite Velocity Research Platform consisting of:</li> </ul> |
| | o EnSite Velocity Research Display Workstation (CE marked) |
| | o EnSite Velocity Research Switch (OEM CE marked) |
| | <ul> <li>EnSite Velocity Research software (not CE marked)</li> <li>Any commercially available Radiofrequency (RF) ablation system</li> </ul> |
| | - Any commercially available irrigated tip RF ablation catheter |
| | (minimum 4 electrodes) |
| Study Population | - Any CE-marked EP diagnostic catheter (minimum 4 electrodes) Patients with persistent AF scheduled to undergo first or second time catheter |
| Study I opulation | ablation with approved standard indication by ESC/EHRA Guidelines |
| Inclusion/Exclusion | Inclusion Criteria |
| Criteria | 1. Age between 18 and 85 years |
| | <ul><li>2. Persistent AF</li><li>3. Ability to provide informed consent for study participation and be willing</li></ul> |
| | and able to comply with study evaluations and follow-up schedule |

| Clinical Investigational Plan Synopsis |
|---|
| Study Name: Substrate-targeted Catheter Ablation to Treat Atrial Fibrillation Ver. 1.0 11MAR2015 |

# **Clinical Investigational Plan Synopsis**

| | Exclusion Criteria | | |
|---|---|---|---|
| | 1. Two or more previous AF ablations | | |
| | 2. Secondary AF | | |
| | 3. Hyperthyroidism | | |
| | 4. Left ventricular ejection fraction <30% | | |
| | 5. NYHA functional class IV | | |
| | 6. Left atrial area > 35 cm <sup>2</sup> | | |
| | 7. Uncorrected severe valvular heart disease | | |
| | 8. Contraindication to anticoagulation | | |
| | 9. Presence of left atrial thrombus | | |
| | 10. Recent (<6 Months) myocardial Infarction or unstable angina or coronary artery by-pass | | |
| | 11. Thoracic surgery for congenital, valvular or aortic disease | | |
| | 12. History of cerebrovascular accidents | | |
| | 13. Pregnancy | | |
| | 14. Significant comorbidities such as cancer, severe renal insufficiency requiring hemodialysis, severe obstructive lung disease, cirrhosis, with a life expectancy less than 2 years | | |
| Data Collection | - Pre-procedure: Data collection per standard clinical practice for | | |
| | patients undergoing AF ablation | | |
| - During-procedure: EnSite Velocity Study Backup DVDs, including 3D geometry of LA, contact maps collected by AFocus II catheter, electrograms, RF lesion locations, marker locations, electrode | | | |
| | | locations, user annotations, events of acute AF termination or | |
| | | | significant CL slowing |
| | Post-procedure: AF recurrence documented by ILR or TT ECG monitoring | | |

Clinical Investigational Plan Synopsis Study Name: Substrate-targeted Catheter Ablation to Treat Atrial Fibrillation Ver. 1.0 11MAR2015

## **Clinical Investigational Plan Synopsis**

#### 1. Study Flow Chart



| Clinical Investigational Plan Synopsis |
|---|
| Study Name: Substrate-targeted Catheter Ablation to Treat Atrial Fibrillation Ver. 1.0 11MAR2015 |

## **Clinical Investigational Plan Synopsis**

### 2. Statistical analysis

In subjects with persistent AF, it is possible to demonstrate a one-year clinical difference among the two therapies with a significance level of 0.5 and a power of 0.80 using a Log-rank test in 38 subjects per group, estimated success of 50% and 80% in the control arm and mapping arm, respectively. The expected difference is based on extensive experience of the operators. Considering 5% drop-out rates, thus a total of 80 subjects will be included and assigned to either treatment group according to a randomization schedule stratified by the previous ablation procedures (none and one previous ablation procedure). Categorical and continuous variables are expressed as absolute and relative frequencies or as mean $\pm$ SD or median (interquartile range [IQR]) as appropriate. Comparisons of continuous variables were done with a Student t-test or the Mann-Whitney U test as appropriate and binomial variables with chi-square or Fisher test. Long-term outcome was assessed, after a single ablation procedure, by Kaplan-Meier method and compared using the log rank test. A 2-tailed probability value of  $\leq$  0.05 was deemed significant. Statistical analyses were conducted using SPSS (SPSS v22, USA).